CLINICAL TRIAL: NCT01988077
Title: Clinical Evaluation of Yervoy in Combination With Adoptive T Cell Transfer for the Treatment of Metastatic Melanoma Patients
Brief Title: Clinical Evaluation of Yervoy in Combination With Adoptive T Cell Transfer for Metastatic Melanoma Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to toxicity of cyclophosphamide
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Jacob Schachter MD,, Head - Ella Institute for Melanoma, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ipilimumab TIL
Record Dates: First submitted 2013-10-24; First posted 2013-11-20 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: A Combination of Adoptive T Cell Therapy and Ipilimumab Could Increase the Proportion of CR Patients, and Durability of Response
MeSH Terms: interventions — Adoptive Transfer; Ipilimumab; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adoptive cell transfer combined with Ipilimumab (Other): Adoptive cell transfer combined with Ipilimumab
  Interventions: Biological: Adoptive cell transfer; Drug: Ipilimumab 5 MG/ML Injection [Yervoy]

INTERVENTIONS:
Biological: Adoptive cell transfer — Adoptive cell transfer
Drug: Ipilimumab 5 MG/ML Injection [Yervoy] — 2 treatments of Ipilimumab before transfer of TIL and 2 treatments of Ipilimumab after TIL

SUMMARY:
A rationally designed combination of adoptive T cell therapy and ipilimumab could strongly increase the proportion of CR patients, as well as the durability of response, as compared to ipilimumab or TIL alone. The investigators hypothesize that the combination of those two important modalities could result in a durable (≥ 1 year) complete response rate of 30% in stage IV melanoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ≥ 18 years of age.
* Measurable metastatic melanoma (defined histologically) with at least one lesion that is resectable for TIL generation:
* Patients with asymptomatic brain metastases are allowed
* Previously treated or untreated unresectable stage III or stage IV melanoma
* Clinical performance status of ECOG 0 or 1.
* Laboratory:

  * ANC ≥ than 1000 k/microL without support of filgrastim
  * WBC > 3000 k/microL
  * Hemoglobin greater than 8.0 g/dL
  * Platelet count greater than 100,000 K/microL
  * Seronegative for HIV, HBV, HCV
  * Serum ALT/AST less than three times the upper limit of normal.
  * Serum creatinine less than or equal to 1.6 mg/dL.
  * Total bilirubin less than or equal to 2 mg/dL, except in patients with Gilbert's syndrome who must have a total bilirubin less than 3 mg/dl.
* An interval of at least 28 days since last oncological treatment to the first ipilimumab course. Palliative radiation therapy outside of the brain or therapeutic radiation to the brain after the patient's condition is stabilized and systemic steroids required for the management of systems due to brain metastases is decreased to the lowest fixed dose possible does not require 28-day waiting period.
* Negative pregnancy test in women of child bearing potentialwithin 72 hours before the start of ipilimumab.
* Willing to practice effective birth control during treatment and for 26 weeks after receiving the last dose of ipilimumab (both women of child bearing potential and men of fathering potential).
* Life expectancy greater than three months.

Exclusion Criteria:

* Failure to meet all of the inclusion criteria.
* Autoimmune disease: Patients with a history of inflammatory bowel disease, including ulcerative colitis and Crohn's Disease, are excluded from this study, as are patients with a history of symptomatic disease (eg, rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [eg, Wegener's Granulomatosis]); motor neuropathy considered of autoimmune origin (e.g. Guillain-Barre Syndrome and Myasthenia Gravis).
* Active concurrent malignant disease, or disease-free for less than 5 years (exception: adequately treated basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix)
* Patients receiving any non-oncology vaccine therapy used for prevention of infectious diseases for up to 4 weeks before or after any dose of ipilimumab with the exception of amantadine and flumadine, will not be eligible for ipilimumab treatment.
* Any underlying medical or psychiatric condition, which in the opinion of the investigator will make the administration of ipilimumab hazardous or obscure the interpretation of AEs, such as a condition associated with frequent diarrhea.
* Active systemic infections, coagulation disorders or other active major medical illnesses:
* Cardiovascular:

  * History of coronary revascularization or ischemic symptoms
  * Clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block
  * Left ventricular EF of 45% or less.
  * Respiratory:
  * Documented FEV1 less than or equal to 70% tested in patients with symptoms of respiratory dysfunction
  * Immune system
  * Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease and AIDS)
  * Hepatitis B and C infection, regardless of the control on antiviral therapy
  * Opportunistic infections
* Any subject who has a life-threatening condition that requires high-dose immunosuppressant(s).
* A history of prior treatment with ipilimumab or prior CD137 agonist or CTLA 4 inhibitor or agonist
* History of severe immediate hypersensitivity reaction to any of the agents used in this study.
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (eg, infectious) illness.
* Women of child-bearing potential:
* Pregnant, breastfeeding, or unwilling or unable to use an acceptable method of contraception to avoid pregnancy for their entire study period and for at least 8 weeks after cessation of study drug

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-10; Primary Completion 2016-05-20 (Actual); Study Completion 2018-10-25 (Actual)

PRIMARY OUTCOMES:
Determine the response rate of the combination of ipilimumab with young TIL protocol and the CR rate of this combination according to modified RECIST 1.1. | October 2017

SECONDARY OUTCOMES:
• Evaluate the toxicity of this treatment regimen. | Follow up for 1 year
  Toxicity will be reported by type and severity according to the National Cancer Institute Common Toxicity Criteria (NCI CTC) version 4.

OTHER OUTCOMES:
Determine duration of response | follow up for 1 year
Determine overall survival | follow up for 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Schachter, Prof., Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba. Medical Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: Undecided
to be decided